CLINICAL TRIAL: NCT06439849
Title: Single Patient Compassionate Use / Expanded Access L-S-Gboxin (Lyophilized Form of S-Gboxin) for the Treatment of Diffuse Midline Glioma, H3 K27/K28-altered (TRIANGLE)
Brief Title: Single Patient Compassionate Use / Expanded Access L-S-Gboxin (Lyophilized Form of S-Gboxin) for the Treatment of Diffuse Midline Glioma
Acronym: TRIANGLE
Status: No longer available | Type: Expanded Access
Sponsor: Petrov, Andrey (Other)
Responsible Party: Sponsor
Other Study IDs: 21DN24S
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: DIPG Brain Tumor; Diffuse Brainstem Glioma; H3 K27M; H3 K28M; GBM
Keywords: S-Gboxin; S-Gboxin (lyophilized form)
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: S-Gboxin — S-Gboxin (lyophilized form of S-Gboxin) for the treatment diffuse midline glioma with H3 K27M / H3 K28M mutation
  Other Names: lyophilized form of S - Gboxin; 3-(2-(((1R,2S,5R)-2-isopropyl-5-methylcyclohexyl)oxy)-2-oxoethyl)-1-methyl-2-(3-(trifluoromethyl)phenyl)-1H-benzo[d]imidazol-3-ium iodide

SUMMARY:
F. 50y.o. 77kg, DS confirmed 18 Nov. 2022 Received treatment: 11 courses of TMZ (240mg) Radiotherapy 30 courses of 1.8Gr (total 54 Gr, TMZ 140 mg on RT). Bevacizumab intravenously -400 mg -0-14-28-42 (December-February 2023). Severe side effects. The attending physician discontinued bevacizumab after 4 courses. In remission for 11 months. According to the results of the MRI dated April 28, 2024, continued growth.

Neurological status is good. Reflexes are not impaired. To date, treatment options have been exhausted. Participation of the patient in Clinical Trials is impossible. As of April 2024, negative dynamics. The patient signed an informed consent agreement. Information on taking L-S-Gboxin (Lyophilisate) as part of a compassionate program - explained.

Written consent of the attending physician for the patient's participation in the Compassion Program (TRIANGLE) with L-S-Gboxi (Lyophilisate) - received.

(medical documentation will be available on clinicaltrials.gov within a month from the date of publication - patient's consent to publish the medical history and examination results has been obtained)

DETAILED DESCRIPTION:
TREATMENT PLAN

Оn days 1 to 3 of treatment, the patient will receive a sublingual form of the lyophilized form of L-S-Gboxin at a dose of 5 mg/kg.

If there is no toxicity, on days 4 to 14 the patient will receive a sublingual form of the lyophilized form of S-Gboxin at a dose of 10 mg/kg.

The first course of treatment is 14 days. On day 20, MRI + PET-CT monitoring is carried out to assess the dynamics of tumor growth. Based on the results of the examination plan, the attending physician and the main investigator make a decision on the continuation of treatment and the duration of the second course of therapy.

ELIGIBILITY:
Inclusion Criteria:

unacceptable for single patient

Exclusion Criteria:

* unacceptable cardiotoxicity
* cerebrospinal fluid dissemination
* systemic infection or viral disease, other associated symptoms that may jeopardize the patient's safety (at the discretion of the treating physician)

Age Groups: Child, Adult, Older Adult

REFERENCES:
- See also: OXPHOS — https://www.nature.com/articles/ncomms4103
- See also: Gboxin — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6655586/
- See also: OXPHOS — https://pubmed.ncbi.nlm.nih.gov/37736880/